CLINICAL TRIAL: NCT03255421
Title: Filling and Emptying Cystometries: a Feasibility and Validation Study in Order to Simplify the Manometric Follow-up of Overactive Detrusor in Neurological Patients Under Anticholinergic or Botulinum Toxin Injections.
Brief Title: Filling and Emptying Cystometries ("Backwards Cystometry"): a Feasibility and Validation Study
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon hospital, Pierre and Marie Curie University
Other Study IDs: P GREEN 01
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: urodynamic; backwards cystometry; reverse cystometry; follow-up
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patients over 18 years old, consulting for lower urinary tract symptoms and performing an urodynamic examination with a cystometry in a tertiary center are included.
  First pressure measurement in the bladder during the classic cystometry. Second measurement of bladder pressures during the bladder emptying.
  Interventions: Other: Pressure measurement

INTERVENTIONS:
Other: Pressure measurement — Observational study No intervention, only fragmenting the emptying of the bladder

SUMMARY:
This study evaluate the feasibility and the accuracy of an emptying cystometry in order to simplify the manometric follow-up of overactive detrusor in neurological patients under anticholinergic or botulinum toxin injections.

DETAILED DESCRIPTION:
Bladder pressure assessment is necessary for the diagnosis, the prognostic assessment and the management of neurogenic bladder. High bladder pressures increase the rate of urological complications and mortality in patients with neurogenic bladder. Thus many treatments are proposed in order to improve bladder compliance and reduce uninhibited detrusor contractions (anticholinergic drugs, botulinum toxin injections, cystoplasty, sacral neuromodulation, beta-3-agonist, posterior tibial nerve stimulation).

Clinical data, symptoms scales, quality of life questionnaires, renal ultrasound, biological tests of renal function and urodynamic studies are used to control the treatment efficacy of neurogenic lower urinary tract dysfunction. Filling cystometry is the usual way to record bladder pressure. Urodynamic techniques using external pressure transducers (microtip, air-filled or fluid-perfused catheters) connected to the patient with fluid-filled lines are recommended. This multichannel cystometry is performed in a specialized department with the inconvenience of delays for appointments and cost of the urodynamic assessment. Moreover, only some parameters are important and are taken in account in the follow-up of these neurogenic bladders: bladder capacity, bladder compliance and maximum detrusor pressure at the end of the filling phase. All these parameters can be recorded with a self-assessment of bladder pressure at home with a very simple device made of 1) a self-intermittent catheter; 2) a three way stopcock; 3) a simple graduated tube. This device has in fact been used in the past to realize cystometries, in particular in the elderly subject. A such device should provide a monitoring in changes in bladder pressure in order to initiate adjustments in treatment sooner than would be achieved when patients are evaluated periodically but less frequently in the neurourology department. The early detection of high bladder pressures may avoid bladder deformation, reflux and upper tract deterioration. Moreover, the home control of appropriate bladder pressure may improve the patients' quality of live by reducing the constraint linked to the time-consuming specialized follow-up.

In this study, the investigators will test a reverse single channel cystometry performed just after a classical filling cystometry during the usual emptying by means of a device allowing serial bladder pressure measurements during the bladder emptying. In case of such a feasibility and a good precision of the reverse cystometry, the manometric follow-up of overactive detrusor in neurological patients under anticholinergic or botulinum toxin injections could be simplified.

The aim of this study is to assess the feasibility and the accuracy of sequential measurements of bladder pressure during the bladder emptying and to compare the evolution of bladder pressures during the emptying phase with the bladder pressures recorded during the filling phase.

Patients over 18 years old, consulting for lower urinary tract symptoms and performing an urodynamic examination with a cystometry in a tertiary center are included.

History, treatment and urodynamics data are recorded. Conventional supine multichannel cystometry with isotonic saline infused at 50ml/min (filling cystometry), conform to the International Continence Society (ICS) recommendations will be performed. At the end of the standard cystometry when the maximum cystometric capacity will be reached, if no micturition was obtained, urodynamic catheter was withdrawn and a CH12 urinary catheter will be introduced in the bladder according to the usual department procedure (usually, this catheter allows to empty the bladder). This catheter will be connected to a three-way stopcock. The second way of the stopcock will permit the emptying into a measuring container, graduated each 50ml. The third way of the stopcock will be connected via a tube extension to a rigid vertical 70cm tube (central venous pressure set) graduated each centimeter. The zero pressure of the vertical tube will be set at the upper edge of the symphysis pubis. For measuring the bladder pressure at the maximum cystometric capacity, the valve will be open between the bladder and the graduated tube, manometric data will be derived by observing the rise of the column of fluid in the centimeter scale tube. This procedure will be repeated every 50ml until bladder full emptying.

The investigators will compared each bladder pressure measures every 50ml during the "backwards cystometry" with each bladder pressure measured every 50ml from the maximum capacity during the filling cystometry.

Primary outcome is the agreement between the two cystometries evaluated using a kappa coefficient.

Secondary outcome is the correlation between the pressures during the two cystometries.

ELIGIBILITY:
Inclusion Criteria:

* Follow in neuro-urology for lower urinary tract symptoms
* Appointment for urodynamic assessment

Exclusion Criteria:

* detrusor overactivity
* micturition during or at the end of the filling cystometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting for an urodynamic assessment in a tertiary center in neuro-urology
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Agreement | 1 Day : during the urodynamic assessment
  Agreement between the two cystometries evaluated using a kappa coefficient.

SECONDARY OUTCOMES:
Correlation | 1 Day : during the urodynamic assessment
  Correlation between the pressures during the two cystometries.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — GREEN GRC-01, Neuro-urology, hôpital Tenon
Locations (1):
- Department of Neuro-urology, Tenon hospital, Paris, France